CLINICAL TRIAL: NCT00485849
Title: An Open Label Pilot Study of Atomoxetine for Attention Deficit and Hyperactive/Impulsive Behavior Problems in Children and Adolescents With Autistic Spectrum Disorders
Brief Title: A Study of Atomoxetine for Attention Deficit and Hyperactive/Impulsive Behaviour Problems in Children With ASD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6639; B4Z-UT-S003
Record Dates: First submitted 2007-06-11; First posted 2007-06-13 (Estimated); Last update posted 2007-06-13 (Estimated); Status verified 2007-06

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride

INTERVENTIONS:
Drug: Atomoxetine Hydrochloride

SUMMARY:
The primary purpose of this study is to evaluate the tolerability and effectiveness of atomoxetine in the treatment of attention problems, hyperactivity, and impulsivity in children with ASD, and secondarily, to evaluate the possible response to atomoxetine on the core symptoms of ASD

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients between the ages of at least 6 years of age and not more than 17 years of age at visit 1
* Autistic Spectrum Disorder (DSM-IV TR) diagnosis of Autistic disorder or Asperger syndrome or PDDNOS
* Clinically significant symptoms of ADHD (i.e. inattention, impulsiveness, and hyperactivity) that have been present for at least six months (for subjects older than 8 years, the onset of symptoms must be before the age of 7 years)
* Medication-free for at least two weeks for all psychotropic medications (four weeks for fluoxetine or depot-neuroleptics)
* Patients must also be able to swallow capsules

Exclusion Criteria:

* Patients who weigh less than 20 kg or greater than 60 kg at visit 2
* DSM-IV TR diagnosis of a Pervasive Developmental Disorder other than Autistic Disorder, PDD-NOS, Asperger's Disorder (e.g. Rett's Disorder, Childhood Disintegrative Disorder)
* Patients who have a history of Bipolar I or II disorder, schizophrenia, psychosis
* Patients who have a current diagnosis of Major Depression (with or without psychotic features), PTSD
* Patients with a history of any seizure disorder (other than febrile seizures) or patients who have taken (or are currently taking) anticonvulsants for seizure control

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2004-02; Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Test whether atomoxetine is effective in reducing symptoms of inattention and overactivity/impulsivity as measured by the AHDHRS-IV-Parent:Inv scale in pediatric outpatients with ASD accompanied by ADHD behavior problems

SECONDARY OUTCOMES:
To assess whether atomoxetine will be effective in reducing symptoms of inattention and overactivity/impulsivity
To assess whether atomoxetine will be effective for improving social functioning and personal sufficiency in children and adolescents with ASD+ADHD
To assess whether atomoxetine has a positive or negative effect on frequently associated symptoms as impulsive aggression, agitation, self-injurious behavior, troublesome repetitive behavior and poor motor coordination
To assess whether atomoxetine has a positive or negative effect on neuropsychological functioning
To assess the overall influence on functioning and burden on the family
To monitor clinical safety and side effects as assessed by adverse events elicited during open-ended questioning

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Groningen, Netherlands

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com